CLINICAL TRIAL: NCT00188682
Title: Optical Transillumination Spectroscopy of Breast Tissue in Pre- and Post-Menopausal Women.
Brief Title: Breast Study to Determine the Ability of Non-Invasive Optical Transillumination Spectroscopy to Predict Breast Density.
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Other Study IDs: UHNREB#00-0081-C; DOD#DAMD17-00-1-0393; UTREB#5507
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2007-11-15 (Estimated); Status verified 2007-11

CONDITIONS: Breast Cancer
Keywords: Optical Transillumination Spectroscopy; Transillumination Breast Spectroscopy; Breast Cancer Risk
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to learn more about the application of transillumination measurements in the determination of breast cancer risk. The goal is to demonstrate a correlation between non-invasive optical transillumination spectroscopy and parenchymal density pattern.

DETAILED DESCRIPTION:
X-ray generated images, such as mammograms, rely on the density of tissue within the breast. Tissue density are believed to be associated with proliferation of stroma and/or epithelium, which result in an increase in water associated light absorption and a decrease in lipid associated light absorption. The amount of density of the breast tissue has been shown to be an indicator of cancer risk. Thus, assessing this breast tissue density is also an important tool in determining breast cancer risk.

Optical transillumination has been shown to give information about tissue composition and tissue density. Unlike x-ray mammography which uses ionizing radiation, optical transillumination uses normal white light and is deemed safe to be used frequently for women of all ages and therefore can be used for those situations where mammography is not an option.

Normal white light is shone into the tissue and the light that leaves the breast on the other side from the source is detected and analyzed. Since the same physiological conditions that contribute to dense breast tissue, as seen in mammography, also will have unique optical signatures.

We will compare the amount of this dense tissue from the mammogram, taken with 12 months, to the density measurements found through the optical procedure. The goal is to be able to duplicate the information from the mammogram using the transillumination technique. All measurements are non-invasive and no blood samples or biopsies are required.

ELIGIBILITY:
Inclusion Criteria:

* Be in good health and able to provide consent
* Be between 35 and 75 years of age
* Have no personal history of breast cancer
* Have had a mammogram at The Marvelle Koffler Breast Centre at Mount Sinai Hospital within the last 12 months

Exclusion Criteria:

* Have had breast biopsy
* Have had breast augmentation or reduction

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort recruited from the Marvelle Koffler Centre at Mount Sinai Hospital (Toronto, Ontario, Canada)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2000-03; Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lothar Lilge, PhD, Principal Investigator — Ontario Cancer Institute, University Health Network, Toronto, Ontario, Canada M5G 2M9; Department of Biophysics and Bioimaging, University of Toronto, Toronto, Ontario, Canada M5G 2M9
Locations (1):
- Ontario Cancer Institute, Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Blyschak K, Simick M, Jong R, Lilge L. Classification of breast tissue density by optical transillumination spectroscopy: optical and physiological effects governing predictive value. Med Phys. 2004 Jun;31(6):1398-414. doi: 10.1118/1.1738191. PMID 15259643
- [Result] Simick MK, Jong R, Wilson B, Lilge L. Non-ionizing near-infrared radiation transillumination spectroscopy for breast tissue density and assessment of breast cancer risk. J Biomed Opt. 2004 Jul-Aug;9(4):794-803. doi: 10.1117/1.1758269. PMID 15250768
- [Result] Simick MK, Lilge L. Optical transillumination spectroscopy to quantify parenchymal tissue density: an indicator for breast cancer risk. Br J Radiol. 2005 Nov;78(935):1009-17. doi: 10.1259/bjr/14696165. PMID 16249602
- [Result] Blackmore KM, Knight JA, Jong R, Lilge L. Assessing breast tissue density by transillumination breast spectroscopy (TIBS): an intermediate indicator of cancer risk. Br J Radiol. 2007 Jul;80(955):545-56. doi: 10.1259/bjr/26858614. Epub 2007 May 30. PMID 17537757